CLINICAL TRIAL: NCT07167784
Title: Ecological Momentary Assessment to Explore Fatigue, Pain, Sleep, Mood and Physical Activity Levels in Patients With Inflammatory Rheumatic Disease. A Pilot Study of Feasibility and Acceptability
Brief Title: Ecological Momentary Assessment and Physical Activity in Patients With Inflammatory Rheumatic Diseases
Acronym: DYNAMIC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: EssaiClinique_DYNAMIC
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis &Amp;Amp;Amp; Other Inflammatory Polyarthropathies; Spondyloarthritis (SpA)
Keywords: Ecological Momentary Assessment; Chronic Inflammatory Rheumatic Diseases; physical activity; fatigue; sleep; pain; actigraphy
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Motor Activity; Fatigue; Pain | interventions — Ecological Momentary Assessment

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ecological Momentary Assessment — Participants will be complete four daily EMA surveys via the Avicenna Research app (morning, 11 a.m., 3 p.m., and evening). Participants will be instructed to complete and submit each survey as soon as they see the app notification. If no response is provided within 15 minutes, a reminder notification will be sent. At the end of the 14-day period, devices will be returned using a prepaid envelope provided by the study team and participants will complete an end-of-study questionnaire to assess the acceptability of the study and will be invited to participate in a debriefing interview with a member of the research team.

SUMMARY:
Chronic inflammatory rheumatic diseases (IRDs), such as rheumatoid arthritis and spondyloarthritis, can cause pain, fatigue, and mobility issues, significantly impacting patients' quality of life. Physical activity is an important part of managing these conditions, as it helps reduce pain, maintain mobility, and prevent complications. However, many patients struggle to stay active due to pain and fatigue. Understanding these challenges better could lead to improved support and interventions.

This study explores a new way to monitor the daily experiences of patients with IRDs using Ecological Momentary Assessment (EMA), a method that collects real-time data through a mobile app. The study will also use actimeters-wearable devices that track physical activity. Over 14 days, participants will answer short surveys on their phone and wear an actimeter to provide insights into how fatigue, pain, mood, and physical activity levels change throughout the day.

Before using this approach in a larger study, we need to make sure it is practical and acceptable for patients. This pilot study will assess whether participants find the mobile app and actimeter easy to use, how often they respond to surveys, and whether frequent reminders affect their willingness to participate. The study will also examine the immediate and delayed effects of different symptoms on physical activity and explore factors that influence patient engagement with the protocol.

By identifying potential barriers and solutions, this research will help refine future studies and improve the way we monitor and support people with IRDs in staying active while managing their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with a confirmed diagnosis of CIRDs, including RA or SpA, established by a rheumatologist, are eligible for inclusion. Participants must be able to understand and consent to the study protocol, be affiliated with a social security system, and have access to a digital device with internet access (e.g., smartphone or tablet).

Non-inclusion Criteria:

* Insufficient proficiency in the French language; legal incapacity or deprivation of liberty; major cognitive impairment incompatible with repeated questionnaire completion (e.g., Alzheimer's disease); pregnant or breastfeeding women, as well as individuals with a history of alcohol or substance abuse, or severe psychiatric disorders that could affect adherence to the protocol or the reliability of collected data, are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with Chronic inflammatory rheumatic diseases (rheumatoid arthritis or spondyloarthritis)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a 14-day smartphone EMA protocol combined with actigraphy | Day 1 to Day 14 after enrollment
  Feasibility will be quantified on five pre-specified indicators:
  (1) attrition rates; measured by the number of participants who withdrew from the study, (2) the number and percentage of data collected from EMA surveys relative to the number of potential assessments, (3) the percentage of surveys that a participant started to complete, relative to the number of potential assessments, (4) time elapsed between the prompt and the start of the response to the survey, (5) adherence to actigraphy (the threshold is at least 21 hours of wear time over 24 hours, for 14 days).
Acceptability of a 14-day EMA protocol combined with actigraphy delivered via a mobile application | Day 1 to Day 14 after enrollment
  Acceptability will be assessed at follow-up using a structured questionnaire and semi-structured interviews. The questionnaire will evaluate participant satisfaction, perceived relevance, ease of use, and daily burden associated with EMA and actigraphy. Each item will be rated on a five-point Likert scale (1 = strongly disagree to 5 = strongly agree). Acceptability at the item level will be defined as ≥70% agreement on positively worded items and ≤30% agreement on negatively worded items. A score ≥3/5 will indicate acceptable validation of an item. In addition, semi-structured interviews will be conducted to explore participant experiences; with consent, sessions will be audio-recorded, transcribed in a non-verbatim format, and analyzed using content analysis to identify recurring themes.

SECONDARY OUTCOMES:
Immediate and Lagged Effects on Physical Activity | Day 1 to Day 14 after enrollment
  To examine the temporal relationships between pain, fatigue, and sleep, considering their reciprocal influences and variations across different times of the day
Immediate and Lagged Effects of Determinants on Physical Activity | Day 1 to Day 14 after enrollment
  To describe both the immediate and lagged effects of these factors on objectively measured physical activity
Adherence and Acceptability of Two Actigraph Devices | Day 1 to Day 14 after enrollment
  To compare adherence to and acceptability of two actigraph devices assessing physical activity, sleep, and sedentary behavior, worn at two different body sites
Patient-Perceived Acceptability | Day 1 to Day 14 after enrollment
  To explore the qualitative determinants of protocol acceptability directly from the patients' perspective

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France, France

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this study will be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available 6 months after publication of the main results and will remain available for 5 years.
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal. Requests should be directed to the study coordinator. After approval of the proposal, data will be shared via a secure repository or direct data transfer agreement.

REFERENCES:
- [Derived] Aymard N, Darmaillacq A, Bailly S, Kechichian A, Baillieul S, Bernardy C, Gastaldi R, Flore P, Baillet A, Mendelson M. Ecological momentary assessment of daily patient-reported outcomes and actigraphy-measured physical activity and sleep in patients with rheumatoid arthritis and spondyloarthritis: a study protocol. BMJ Open. 2026 Feb 10;16(2):e113370. doi: 10.1136/bmjopen-2025-113370. PMID 41667166